CLINICAL TRIAL: NCT03004755
Title: The PEACE (Posthumous Evaluation of Advanced Cancer Environment) Study
Acronym: PEACE
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Other Study IDs: UCL/13/0165
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Solid Tumor, Adult; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Tissue and Organ Harvesting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Tissue Harvest

SUMMARY:
Historically, cancer research has been limited by sample acquisition in late stage disease, often restricted to single sites of disease with limited parallel clinical data collection in terms of prior therapy exposure. The PEACE study is intended to facilitate tissue donation from multiple tumour sites in the post-mortem setting and enable future research using samples collected at post-mortem within different disciplines related to cancer research.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Confirmed diagnosis of any form of solid malignancy with metastatic disease (where the site of origin is known or unknown), with the exception of primary brain tumour in which there may not be evidence of metastatic disease
* Oral and written informed consent from patient to enter the study and to undergo tumour harvesting after death or informed consent from a person in a qualifying relationship after the patient has died.

Exclusion Criteria:

* Medical or psychiatric condition that would preclude informed consent
* History of intravenous drug abuse within the last 5 years
* History of known high-risk infections (e.g. HIV/AIDS-positive, hepatitis B/C, tuberculosis and Creutzfeldt-Jacob disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Solid tumour malignancy with metastatic disease
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-03; Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Perform 500 post mortems | 5 years

CONTACTS AND LOCATIONS:
Locations (9):
- United Kingdom (9):
  - Heart of England NHS Foundation Trust, Birmingham
  - Cambridge University NHS Trust, Cambridge
  - Greater Glasgow Health Board, Glasgow
  - University Hospitals of Leicester NHS Trust, Leicester
  - Guy's and St Thomas NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Trust, Oxford

REFERENCES:
- [Derived] Turajlic S, Xu H, Litchfield K, Rowan A, Chambers T, Lopez JI, Nicol D, O'Brien T, Larkin J, Horswell S, Stares M, Au L, Jamal-Hanjani M, Challacombe B, Chandra A, Hazell S, Eichler-Jonsson C, Soultati A, Chowdhury S, Rudman S, Lynch J, Fernando A, Stamp G, Nye E, Jabbar F, Spain L, Lall S, Guarch R, Falzon M, Proctor I, Pickering L, Gore M, Watkins TBK, Ward S, Stewart A, DiNatale R, Becerra MF, Reznik E, Hsieh JJ, Richmond TA, Mayhew GF, Hill SM, McNally CD, Jones C, Rosenbaum H, Stanislaw S, Burgess DL, Alexander NR, Swanton C; PEACE; TRACERx Renal Consortium. Tracking Cancer Evolution Reveals Constrained Routes to Metastases: TRACERx Renal. Cell. 2018 Apr 19;173(3):581-594.e12. doi: 10.1016/j.cell.2018.03.057. Epub 2018 Apr 12. PMID 29656895
- [Derived] Abbosh C, Birkbak NJ, Wilson GA, Jamal-Hanjani M, Constantin T, Salari R, Le Quesne J, Moore DA, Veeriah S, Rosenthal R, Marafioti T, Kirkizlar E, Watkins TBK, McGranahan N, Ward S, Martinson L, Riley J, Fraioli F, Al Bakir M, Gronroos E, Zambrana F, Endozo R, Bi WL, Fennessy FM, Sponer N, Johnson D, Laycock J, Shafi S, Czyzewska-Khan J, Rowan A, Chambers T, Matthews N, Turajlic S, Hiley C, Lee SM, Forster MD, Ahmad T, Falzon M, Borg E, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Hafez D, Naik A, Ganguly A, Kareht S, Shah R, Joseph L, Marie Quinn A, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Oukrif D, Akarca AU, Hartley JA, Lowe HL, Lock S, Iles N, Bell H, Ngai Y, Elgar G, Szallasi Z, Schwarz RF, Herrero J, Stewart A, Quezada SA, Peggs KS, Van Loo P, Dive C, Lin CJ, Rabinowitz M, Aerts HJWL, Hackshaw A, Shaw JA, Zimmermann BG; TRACERx consortium; PEACE consortium; Swanton C. Phylogenetic ctDNA analysis depicts early-stage lung cancer evolution. Nature. 2017 Apr 26;545(7655):446-451. doi: 10.1038/nature22364. PMID 28445469